CLINICAL TRIAL: NCT07104266
Title: Determine Whether Administering Celecoxib During Radiotherapy Can Reduce the Risk of Recurrence of Triple-negative Breast Cancer. Pilot Study
Brief Title: Triple Negative Breast Cancer and Celecoxib. Pilot Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Benoit Paquette, Professor, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TNBC2025-5681
Record Dates: First submitted 2025-07-17; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Triple-Negative Breast Cancer
Keywords: Triple-Negative Breast Cancer; cytokines; Celecoxib
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Celecoxib; Drug Therapy; Radiotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): One capsule placebo after breakfast and one after supper, starting 7 days before radiotherapy and ending 14 days after radiotherapy.
  Interventions: Drug: Placebo
- Celecoxib (celebrex) (Experimental): One capsule celecoxib (100 mg) after breakfast and one after supper, starting 7 days before radiotherapy and ending 14 days after radiotherapy.
  Interventions: Drug: Celecoxib (Celebrex)

INTERVENTIONS:
Drug: Celecoxib (Celebrex) — The participants will take one capsule celecoxib (100 mg) or placebo after breakfast and one after supper, starting 7 days before radiotherapy and ending 14 days after radiotherapy.
  Other Names: Chemotherapy, radiotherapy
  Arms: Celecoxib (celebrex)
Drug: Placebo — Participants will take one capsule of placebo after breakfast and one after supper, starting 7 days before radiotherapy and ending 14 days after radiotherapy.
  Other Names: Chemotherapy, radiotherapy
  Arms: Placebo

SUMMARY:
Relapses occur in 20 to 30% of patients with early-stage triple-negative breast cancer (TNBC), which is characterized by the absence of three receptors: the estrogen receptor (ER), progesterone receptor (PR) and human epidermal growth factor receptor 2 (HER-2). Radiotherapy (RT) can increase or decrease, depending on the patient, the level of cytokines that promote metastasis development. To help prevent the development of metastasis, the cyclooxygenase-2 (COX-2) inhibitor celecoxib will be administered during RT. This treatment aims to prevent RT-induced cytokine increases and, ultimately, improve patient prognosis.

The primary objective of this pilot study is to assess the feasibility of recruiting participants and implementing the study steps, with the intention of conducting a large-scale study in the future. The secondary objective is to evaluate celecoxib ability to inhibit the RT-induced stimulation of cytokines associated with metastasis development. This will be assessed by comparing the levels of these cytokines in plasma samples collected before, during, and after RT. In the exploratory objective, TNBC cells will be incubated in vitro with these plasma samples to determine whether administering celecoxib during RT can prevent increased cancer cell invasion and metastasis formation in mice.

DETAILED DESCRIPTION:
Adults with non-metastatic TNBC will be recruited. The overall aim is to determine whether administering celecoxib during RT could reduce the risk of cancer recurrence. The hypothesis is that celecoxib will block the increase in cytokines, induced by RT, that are known to promote cancer cell invasion and metastasis. The primary objective of this pilot study is to assess the feasibility of recruiting participants and implementing the study steps, with the intention of conducting a large-scale study in the future.

Thirty participants will be recruited and randomized: fifteen will receive celecoxib, and fifteen will receive a placebo. Participants who take a COX-2 inhibitor for other medical indications or medications such as ibuprofen will be excluded.

Participants are recruited after chemotherapy and removal of the tumor by partial mastectomy. They take one capsule celecoxib (100 mg) or placebo after breakfast and one after supper, starting 7 days before RT and ending 14 days after RT. RT will consist of 26 Gy in 5 fractions or 40 Gy in 15 fractions if participants are under 50 years old with lymph node positivity. According to the RT plan, celecoxib will be taken for no longer than 40 days. In a logbook, participants will report when they take celecoxib and if they experience discomfort, such as skin rashes, headaches, or dizziness. Participant follow-up will last 5 years after treatment, according to clinical guidelines, which include a clinical examination and a mammogram every year. If breast density is categorized as D (extremely dense), an MRI will be performed in alternating years with the mammogram. A CT or PET scan will be conducted if symptoms such as bone pain are present. The date corresponding to the detection of a local or distant recurrence will be recorded in the participant's file to determine whether taking celecoxib could reduce the risk of regional or distant recurrence.

The secondary objective is to determine whether taking celecoxib will prevent the increase in cytokines induced by RT, some of which are known to stimulate the invasion capacity of cancer cells and the formation of metastases. This will be determined by collecting plasma samples at four time points: 1) the day before the start of taking celecoxib or placebo, which corresponds to 7 days before starting RT, 2) the day of the start of RT and just before administering the 1st fraction of radiation, 3) after the 4th fraction of radiation, and 4) 14 days after the end of RT and stopping taking celecoxib or placebo. During the blood draw, participants will be questioned by the research nurse to ensure that celecoxib is well tolerated. The impact of celecoxib on changes in cytokines will be determined using laser bead multiplexing.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age: 18 years or older
* Tumor stage: Early
* TNBC status confirmed by pathology
* Regional lymph node N0 to N3
* No evidence of distant metastasis
* Primary tumor removed by conservative surgery with negative margins

Exclusion Criteria:

Participants will be excluded if they have experienced any of the following conditions in the last six months:

* Stomach ulcer
* Kidney disease: Glomerular filtration rate lower than 50 mL/min
* Liver disease: Aspartate aminotransferase / Alanine aminotransferase - 3 times the upper limit of normal, Bilirubine - 2 times the upper limit of normal, INR - 1.3 times the upper limit of normal, Cirrhose Child-Pugh B or more
* Congestive heart failure: Left ventricular ejection fraction lower than 50%
* Participants taking an NSAID for another medical condition or as needed before starting their radiotherapy treatment.

Participants who have demonstrated:

* Hypersensitivity to celecoxib
* A history of allergic reactions to sulfonamides
* A history of asthma attacks, urticaria, or allergic reactions after taking acetylsalicylic acid or another nonsteroidal anti-inflammatory drug
* The presence of inflammatory bowel disease
* Proven hyperkalemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-04 (Estimated); Primary Completion 2028-08-04 (Estimated); Study Completion 2032-08-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants needed to assess the reduction in recurrence rate by administering celecoxid during radiotherapy | Up to 36 months
  This pilot study aims to assess the feasibility of recruiting participants to take celecoxib during radiotherapy and to estimate the sample size required to obtain statistically significant results (p-value ≤ 0.05), which will be the subject of a subsequent larger-scale study. A reduction of 20% of recurrence rate 3 years post-radiotherapy will be used to estimate the sample size.

SECONDARY OUTCOMES:
Determine the ability of celecoxib to prevent the stimulation of cytokine levels induced by radiotherapy. | Up to 45 days
  The secondary objective is to evaluate the ability of celecoxib to inhibit the radiotherapy-induced elevation of cytokines associated with cancer cell invasion and metastasis development. This will be determined by quantifying and comparing the level of cytokines in plasma samples collected from 30 participants at 4 times: 1) The day before the start of taking celecoxib or placebo, which corresponds to 7 days before starting radiotherapy, 2) the day of the start of radiotherapy and just before administering the 1st fraction of radiation, 3) after the 4th fraction of radiation, and 4) 14 days after the end of radiotherapy and stopping taking celecoxib or placebo.

OTHER OUTCOMES:
Ability of celecoxib to prevent radiotherapy-stimulation of cancer cell invasion | Up to 45 days
  Three triple-negative breast cancer cell lines will be incubated with the four plasma samples collected from each participant. After incubation with these plasma samples, the invasiveness of the cancer cells will be measured in vitro using invasion chambers. In participants receiving a placebo, the plasma collected during radiotherapy is expected to increase the invasiveness of triple-negative breast cancer cells, compared to the two plasma samples collected before radiotherapy.
  By preventing the radiotherapy-induced increase in cytokines associated with cancer cell invasion, celecoxib is expected to block radiotherapy-induced enhancement of cancer cell invasion. Plasma samples collected 14 days after radiotherapy will help determine whether celecoxib's protective effect persists over time.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Paquette, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Faculty of medicine and health sciences, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Age, tumor diameter, stage, chemotherapy and radiotherapy plans, Ki-67 status, administration of pembrolizumab, quantification of cytokine levels in plasma, and relapse 5-years post-treatment
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: August 2025 to August 2032
Access Criteria: Clinicians and basic researchers may request study data from the principal investigator. Participants' clinical data, such as age and disease stage, as well as data collected during the study, will be made available.

DOCUMENTS (1):
  • Study Protocol (2025-07-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT07104266/Prot_000.pdf